CLINICAL TRIAL: NCT03147391
Title: Percutaneous Left Atrial Appendage Closure Using the LAmbre Device in Patients With Atrial Fibrillation: a Single-center, Retrospective, Long-term Real-world Study
Brief Title: Left Atrial Appendage Closure With the LAmbre
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ya-Wei Xu, Director, Head of Cardiology, Principal Investigator, Shanghai 10th People's Hospital
Other Study IDs: LAmbre in real world
Record Dates: First submitted 2017-04-09; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Closure; Stroke
Keywords: Atrial Fibrillation; Left Atrial Appendage Closure; LAmbre device; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LAA closure with LAmbre: The patients with atrial fibrillation who received left atrial appendage (LAA) closure using the LAmbre device in our center from April 2014 to November 2015.
  Interventions: Device: LAA closure with LAmbre

INTERVENTIONS:
Device: LAA closure with LAmbre — Percutaneous Left Atrial Appendage Closure Using the LAmbre Device in Patients With Atrial Fibrillation

SUMMARY:
The study was to retrospectively analyse the efficacy and safety of LAA closure using the LAmbre in our center from April 2014 to November 2015.

DETAILED DESCRIPTION:
The study was to retrospectively analyse the efficacy and safety of percutaneous left atrial appendage (LAA) closure using the LAmbre (Lifetech Scientific Co., Ltd., Shenzhen, China) in our center from April 2014 to November 2015. 89.4% has finished the 12-month esophageal ecllocardiogrhy (TEE) examination. The average followup was 2-years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years of age;
2. Chronic atrial fibrillation ≥3 months; paroxysmal, persistent or permanent non-valvular AF;
3. CHADS2-VAS score 2 or higher;
4. Patient can understand the trial purpose, voluntarily join this clinical trial with informed consent;
5. Patient voluntarily completes the follow-up and follow-up inspection in accordance with the clinical trials process.

Exclusion Criteria:

• A. Clinical exclusion criteria

1. Presence of rheumatic, degenerative or congenital valvular heart diseases,
2. The diameter of left atrial ≥65 mm;
3. LAA size < 12mm or > 30 mm
4. Left atrium has been removed;
5. Heart transplantation patients;
6. Symptomatic patients with carotid artery disease (such as carotid stenosis ≥ 50%);
7. Acute myocardial infarction or unstable angina;
8. Decompensated heart failure (New York Heart Association functional class III-IV);
9. Recent myocardial infarction (< 3 months);
10. Patients with an atrial septal defect or received an atrial septal occluder. The patient has an ablation procedure planned within 30 days of potential LAmbre Occluder implant
11. The patient has a planned cardioversion 30 days post implant of the LAmbre Occluder
12. Patient who after artificial mechanical heart valve replacement operation;
13. Uncontrolled Heart rate ≥ 110 beats / min17) History stroke or TIA within 30 days;
14. Presence of complex aortic plaque(4mm) in ascending aorta;
15. Cardiac tumors or other malignancy with estimated life expectancy u less than 2 years;
16. Have thrombocytopenia (platelet 《105 / μl) or anemia（Hb<10g/dl）;
17. Women who is pregnancy or plan to pregnancy during the trial period;
18. Presence of active sepsis or endocarditis;
19. Patient participated in the other trials;
20. The investigators expect the patient not be able to complete the trial according to requirements.

B. Esophageal ultrasonic exclusion criteria

1. LVEF≤30%;
2. Presence of left atrial appendage thrombus;
3. High risk PFO patients(presence of atrial septal aneurysm);
4. Have obvious mitral valve stenosis (the area of mitral valve≤ 2 cm2);
5. Have obvious and unexplained pericardial effusion(≥4 cm2).
6. Presence of complex aortic plague(≥4 mm) in ascending aorta.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The aim of this retrospective study was to evaluate the long-term follow-up results associated with left atrial appendage closure (LAAC) with the LAmbre (Lifetech Scientific Corp., Shenzhen, China) in patients with nonvalvular atrial fibrillation (NVAF).
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Ischemic stroke | up to 5 years
  Ischemic stroke

SECONDARY OUTCOMES:
The composite safety and efficacy end-points | up to 5 years
  all-cause death, stroke, major bleeding, thromboembolism, device related severe complications
Successful sealing of the LAA | up to 5 years
  successful sealing around the device at the LAA orifice (residual jet flow of < 5 mm) as measured by transesophageal echocardiogram (TEE) at 6 months after device implantation

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, MD, PHD, Study Director — Shanghai 10th People's Hospital

IPD SHARING:
Plan to Share IPD: No